CLINICAL TRIAL: NCT00855790
Title: Comparison of Two Types of Biopsy Forceps for Obtaining Cold Biopsy Polypectomy for Small Sessile Colorectal Polyps Less Than 6 mm in Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: colon polypectomy
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Colorectal Polyps
Keywords: evaluate the effectiveness of one bite polypectomy with the RJ3 biopsy forcep versus the RJ4 biopsy forcep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RJ3 Biopsy Forcep (Active Comparator): use of RJ3 Biopsy forcep for the polypectomy
  Interventions: Other: evaluate the effectiveness of the RJ4 biopsy forcep versus the RJ3 biopsy forcep
- RJ4 Biopsey Forcep (Active Comparator): Use of RJ$ biopsy forcep for polypectomy
  Interventions: Other: evaluate the effectiveness of the RJ4 biopsy forcep versus the RJ3 biopsy forcep

INTERVENTIONS:
Other: evaluate the effectiveness of the RJ4 biopsy forcep versus the RJ3 biopsy forcep — Use of either the RJ3 or RJ4 biopsy forcep for colon polypectomy. will evaluate the effectiveness of removal of polyps less than 6 mm.

SUMMARY:
The purpose of this study is to evaluate the efficacy of the new RJ4 compare with the standard RJ3 biopsy forceps for performing polypectomy for small colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

* colon polyps less than 6 mm

Exclusion Criteria:

* no colon polyps

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Complete endoscopic (visual) eradication of the polyp with the first forceps bite | one year

SECONDARY OUTCOMES:
Number of bites to completely visually eradicate the polyp if the polyp was not fully eradicated with the first forceps bite | one year
Complete pathologic eradication of the polyp on the first forceps bite. | one year
Correlate endoscopic with pathologic eradication | one year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Draganov, MD, Principal Investigator — University of Florida
Locations (1):
- Shands Endocopy Center, Gainesville, Florida, United States

REFERENCES:
- [Derived] Draganov PV, Chang MN, Alkhasawneh A, Dixon LR, Lieb J, Moshiree B, Polyak S, Sultan S, Collins D, Suman A, Valentine JF, Wagh MS, Habashi SL, Forsmark CE. Randomized, controlled trial of standard, large-capacity versus jumbo biopsy forceps for polypectomy of small, sessile, colorectal polyps. Gastrointest Endosc. 2012 Jan;75(1):118-26. doi: 10.1016/j.gie.2011.08.019. PMID 22196811